CLINICAL TRIAL: NCT03766724
Title: A Randomized, Open-label, Multiple-dose, Crossover Study to Investigate the Pharmacokinetic and Pharmacodynamic Drug-Drug Interaction of Evogliptin 5 mg and Empagliflozin 25 mg or Dapagliflozin 10 mg After Oral Administration in Healthy Male Adults
Brief Title: Pharmacokinetic and Pharmacodynamic Drug-Drug Interaction of Evogliptin and Empagliflozin or Dapagliflozin in Healthy Male Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: DA1229_DIS_I
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — empagliflozin; dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): Evogliptin→Evogliptin+Empagliflozin→Empagliflozin
  Interventions: Drug: Evogliptin→Evogliptin+Empagliflozin→Empagliflozin
- Group B (Experimental): Empagliflozin→Evogliptin→Evogliptin+Empagliflozin
  Interventions: Drug: Empagliflozin→Evogliptin→Evogliptin+Empagliflozin
- Group C (Experimental): Evogliptin→Evogliptin+Dapagliflozin→Dapagliflozin
  Interventions: Drug: Evogliptin→Evogliptin+Dapagliflozin→Dapagliflozin
- Group D (Experimental): Dapagliflozin→Evogliptin→Evogliptin+Dapagliflozin
  Interventions: Drug: Dapagliflozin→Evogliptin→Evogliptin+Dapagliflozin

INTERVENTIONS:
Drug: Evogliptin→Evogliptin+Empagliflozin→Empagliflozin — Evogliptin : Evogliptin 5mg QD, Evogliptin+Empagliflozin : Evogliptin 5mg QD + Empagliflozin 25mg QD, Empagliflozin : Empagliflozin 25mg QD
  Other Names: Suganon; Jardiance
  Arms: Group A
Drug: Empagliflozin→Evogliptin→Evogliptin+Empagliflozin — Empagliflozin : Empagliflozin 25mg QD, Evogliptin : Evogliptin 5mg QD, Evogliptin+Empagliflozin : Evogliptin 5mg QD + Empagliflozin 25mg QD
  Other Names: Suganon; Jardiance
  Arms: Group B
Drug: Evogliptin→Evogliptin+Dapagliflozin→Dapagliflozin — Evogliptin : Evogliptin 5mg QD, Evogliptin+Dapagliflozin : Evogliptin 5mg QD + Dapagliflozin 10mg QD, Dapagliflozin : Dapagliflozin 10mg QD
  Other Names: Suganon; Forxiga
  Arms: Group C
Drug: Dapagliflozin→Evogliptin→Evogliptin+Dapagliflozin — Dapagliflozin : Dapagliflozin 10mg QD, Evogliptin : Evogliptin 5mg QD, Evogliptin+Dapagliflozin : Evogliptin 5mg QD + Dapagliflozin 10mg QD
  Other Names: Suganon; Forxiga
  Arms: Group D

SUMMARY:
A Randomized, Open-label, Multiple-dose, Crossover Study to Investigate the Pharmacokinetic and Pharmacodynamic Drug-Drug Interaction of Evogliptin 5 mg and Empagliflozin 25 mg or Dapagliflozin 10 mg after Oral Administration in Healthy Male Adults

ELIGIBILITY:
Inclusion Criteria:

* Health Male Volunteers (Age : 19~55 years)
* Body Weight≥55kg, 18.5≤BMI<25.0

Exclusion Criteria:

* galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
* Allergy or Drug hypersensitivity
* Clinically significant Medical History
* AST, ALT > Upper Normal Range*1.25, eGFR<60mL/min/1.73㎡
* Drink during clinical trial period
* Smoking during clinical trial period
* Grapefruit/Caffeine intake during clinical trial period
* No Contraception

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2018-11-22 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-18 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss | 4 weeks
  area under the concentration-time curve
Cmax,ss | 4 weeks
  maximum serum concentration

CONTACTS AND LOCATIONS:
Overall Officials: Min soo Park, M.D., Ph.D., Principal Investigator — Clinical Trial Center, Severance Hospital
Locations (1):
- Clinical Trials Center, Severance Hospital, Seoul, South Korea